CLINICAL TRIAL: NCT00763867
Title: Phosphodiesterase-5 Inhibition to Improve Clinical Status and Exercise Capacity in Diastolic Heart Failure (RELAX)
Brief Title: Evaluating the Effectiveness of Sildenafil at Improving Health Outcomes and Exercise Ability in People With Diastolic Heart Failure (The RELAX Study)
Acronym: RELAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00018007; U01HL084904 (NIH); U01HL084904-01 (NIH); 521
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Heart Failure, Diastolic; Decompensated Heart Failure; Sildenafil; Exercise Capacity
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — Sugars; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 20 mg three tid for 12 weeks followed by 60 mg tid for 12 weeks
  Interventions: Drug: Placebo
- Sildenafil (Experimental): Sildenafil 20 mg three tid for 12 weeks followed by 60 mg tid for 12 weeks
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Placebo
  Other Names: Sugar pill to mimic Sildenafil
  Arms: Placebo
Drug: Sildenafil
  Other Names: Active Sildenafil
  Arms: Sildenafil

SUMMARY:
Diastolic heart failure (DHF), which affects older individuals and women at a disproportionate rate, is a condition that can lead to shortness of breath and fluid build-up in the lungs. This study will evaluate the effectiveness of the medication sildenafil at improving exercise ability and health outcomes in people with DHF.

DETAILED DESCRIPTION:
DHF is a condition in which one of the chambers of the heart, the left ventricle, loses its ability to relax completely because the muscle has become too stiff. When this occurs, the heart is unable to properly fill with blood, which can lead to decreased blood circulation. People with DHF may experience shortness of breath and pulmonary congestion, which is an abnormal build-up of fluid in the lungs. Current treatment for DHF includes guidelines/recommendations to lower blood pressure, stop smoking, and lose weight, but there are no medications available to specifically treat DHF. Sildenafil, commonly known as Revatio or Viagra, is a medication that increases the supply of blood to the lungs and reduces the workload of the heart. Preliminary studies have shown that sildenafil may be beneficial at improving heart and lung function in people with DHF, but more research is needed to confirm these findings. The purpose of this study is to determine if sildenafil can improve exercise ability and health outcomes in people with DHF.

This 24-week study will enroll people with DHF. Participants will be randomly assigned to receive either sildenafil or placebo three times a day for 24 weeks. Participants will attend study visits at baseline and Weeks 1, 4, 12, 13, and 24. At most study visits, the following procedures will occur: physical exam, medical history review, questionnaires, blood collection, 6-minute walk test to measure endurance, and an exercise test. At baseline and Week 24, participants will also undergo an electrocardiogram, which will measure the electrical activity of the heart, and a cardiac magnetic resonance imaging (MRI) procedure and an echocardiogram, which will both obtain pictures of the heart. At Weeks 3, 8, 16, and 20, study researchers will call participants to collect health information.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of heart failure with current New York Heart Association (NYHA) Class II-IV symptoms
* Has experienced at least one of the following in the 12 months before study entry:

  * Hospitalization for decompensated heart failure
  * Acute treatment with intravenous loop diuretic or hemofiltration
  * Mean pulmonary capillary wedge pressure greater than 15 mm Hg or left ventricular end diastolic pressure (LVEDP) greater than 18 mm Hg at catheterization for dyspnea
  * Long term treatment with a loop diuretic and chronic diastolic dysfunction on echocardiography, as determined by left atrial enlargement
* Left ventricular ejection fraction greater than or equal to 50%, as determined by a clinical echocardiogram or ventriculogram in the 12 months before study entry
* Receiving stable medical therapy in the 30 days before study entry, as determined by no addition or removal of angiotensin converting enzyme inhibitor (ACE), angiotensin receptor blocker (ARB), beta-blockers, or calcium channel blockers (CCB) and no change in dosage of ACE, ARBs, beta-blockers, or CCBs of more than 100%

Exclusion Criteria:

* Has a neuromuscular, orthopedic, or other non-cardiac condition that prevents individual from exercise testing on a bicycle ergometer or from walking in a hallway
* Non-cardiac condition that limits life expectancy to less than 1 year at the time of study entry, based on the judgment of the physician
* Current or anticipated future need for nitrate therapy
* Valve disease (i.e., greater than mild aortic or mitral stenosis; greater than moderate aortic or mitral regurgitation)
* Hypertrophic cardiomyopathy
* Infiltrative or inflammatory myocardial disease (e.g., amyloid, sarcoid)
* Pericardial disease
* Primary pulmonary arteriopathy
* Has experienced a heart attack or unstable angina, or has undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) in the 60 days before study entry, or requires either PTCA or CABG at the time of study entry
* Other clinically important causes of dyspnea, such as morbid obesity or significant lung disease, as defined by clinical judgment or use of steroids or oxygen for lung disease
* Systolic blood pressure less than 110 mm Hg or greater than 180 mm Hg
* Diastolic blood pressure less than 40 mm Hg or greater than 100 mm Hg
* Resting heart rate (HR) greater than 100 bpm
* History of reduced ejection fraction (less than 50%)
* Implanted metallic device that will interfere with MRI examination (in people without atrial fibrillation)
* Severe kidney dysfunction (estimated glomerular filtration rate [GFR] less than 20 ml/min/1.73m2 by modified modification of diet in renal disease [MDRD] equation)
* Pregnant or not using an effective form of contraception
* Hemoglobin level of less than 10 g/dL
* Taking alpha antagonists or cytochrome P450 3A4 inhibitors (e.g., ketoconazole, itraconazole, erythromycin, saquinavir, cimetidine, or serum protease inhibitors for HIV)
* Retinitis pigmentosa, previous diagnosis of nonischemic optic neuropathy, untreated proliferative retinopathy, or unexplained visual disturbance
* Sickle cell anemia, multiple myeloma, leukemia, or penile deformities that increase the risk for priapism (e.g., angulation, cavernosal fibrosis, Peyronie's disease)
* Severe liver disease (aspartate aminotransferase [AST] level greater than three times the normal limit, alkaline phosphatase or bilirubin greater than two times the normal limit)
* In being consistent with American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, people with dyspnea and risk factors for coronary artery disease should have had a stress test and those people with a clinically indicated stress test demonstrating significant ischemia in the 1 year before study entry will be excluded.
* Listed for heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L. Lee, PhD, Principal Investigator — Duke Clinical Research Institute; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (10):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Morehouse School of Medicine, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minnesota Heart Failure Network, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Murray, Utah
  - University of Vermont - Fletcher Allen Health Care, Burlington, Vermont
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Redfield MM, Chen HH, Borlaug BA, Semigran MJ, Lee KL, Lewis G, LeWinter MM, Rouleau JL, Bull DA, Mann DL, Deswal A, Stevenson LW, Givertz MM, Ofili EO, O'Connor CM, Felker GM, Goldsmith SR, Bart BA, McNulty SE, Ibarra JC, Lin G, Oh JK, Patel MR, Kim RJ, Tracy RP, Velazquez EJ, Anstrom KJ, Hernandez AF, Mascette AM, Braunwald E; RELAX Trial. Effect of phosphodiesterase-5 inhibition on exercise capacity and clinical status in heart failure with preserved ejection fraction: a randomized clinical trial. JAMA. 2013 Mar 27;309(12):1268-77. doi: 10.1001/jama.2013.2024. PMID 23478662
- [Derived] Chiu L, Agrawal V, Armstrong D, Brittain E, Collins S, Hemnes AR, Hill JA, Lindenfeld J, Shah SJ, Stevenson LW, Wang TJ, Gupta DK. Correlates of Plasma NT-proBNP/Cyclic GMP Ratio in Heart Failure With Preserved Ejection Fraction: An Analysis of the RELAX Trial. J Am Heart Assoc. 2024 Apr 2;13(7):e031796. doi: 10.1161/JAHA.123.031796. Epub 2024 Mar 27. PMID 38533961
- [Derived] Bevan GH, Rana M, Al-Furaih N, Dalton J, Zidar DA, Al-Kindi SG. Anisocytosis is associated with myocardial fibrosis and exercise capacity in heart failure with preserved ejection fraction. Heart Lung. 2022 Jul-Aug;54:68-73. doi: 10.1016/j.hrtlng.2022.03.013. Epub 2022 Mar 28. PMID 35358904
- [Derived] Reddy YNV, Rikhi A, Obokata M, Shah SJ, Lewis GD, AbouEzzedine OF, Dunlay S, McNulty S, Chakraborty H, Stevenson LW, Redfield MM, Borlaug BA. Quality of life in heart failure with preserved ejection fraction: importance of obesity, functional capacity, and physical inactivity. Eur J Heart Fail. 2020 Jun;22(6):1009-1018. doi: 10.1002/ejhf.1788. Epub 2020 Mar 9. PMID 32150314
- [Derived] Fudim M, Kelly JP, Jones AD, AbouEzzeddine OF, Ambrosy AP, Greene SJ, Reddy YNV, Anstrom KJ, Alhanti B, Lewis GD, Hernandez AF, Felker GM. Are existing and emerging biomarkers associated with cardiorespiratory fitness in patients with chronic heart failure? Am Heart J. 2020 Feb;220:97-107. doi: 10.1016/j.ahj.2019.11.006. Epub 2019 Nov 16. PMID 31805424
- [Derived] Reddy YNV, Lewis GD, Shah SJ, Obokata M, Abou-Ezzedine OF, Fudim M, Sun JL, Chakraborty H, McNulty S, LeWinter MM, Mann DL, Stevenson LW, Redfield MM, Borlaug BA. Characterization of the Obese Phenotype of Heart Failure With Preserved Ejection Fraction: A RELAX Trial Ancillary Study. Mayo Clin Proc. 2019 Jul;94(7):1199-1209. doi: 10.1016/j.mayocp.2018.11.037. PMID 31272568
- [Derived] AbouEzzeddine OF, McKie PM, Dunlay SM, Stevens SR, Felker GM, Borlaug BA, Chen HH, Tracy RP, Braunwald E, Redfield MM. Suppression of Tumorigenicity 2 in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2017 Feb 18;6(2):e004382. doi: 10.1161/JAHA.116.004382. PMID 28214792
- [Derived] DeVore AD, McNulty S, Alenezi F, Ersboll M, Vader JM, Oh JK, Lin G, Redfield MM, Lewis G, Semigran MJ, Anstrom KJ, Hernandez AF, Velazquez EJ. Impaired left ventricular global longitudinal strain in patients with heart failure with preserved ejection fraction: insights from the RELAX trial. Eur J Heart Fail. 2017 Jul;19(7):893-900. doi: 10.1002/ejhf.754. Epub 2017 Feb 14. PMID 28194841
- [Derived] Hussain I, Mohammed SF, Forfia PR, Lewis GD, Borlaug BA, Gallup DS, Redfield MM. Impaired Right Ventricular-Pulmonary Arterial Coupling and Effect of Sildenafil in Heart Failure With Preserved Ejection Fraction: An Ancillary Analysis From the Phosphodiesterase-5 Inhibition to Improve Clinical Status And Exercise Capacity in Diastolic Heart Failure (RELAX) Trial. Circ Heart Fail. 2016 Apr;9(4):e002729. doi: 10.1161/CIRCHEARTFAILURE.115.002729. PMID 27072860
- [Derived] Lindman BR, Davila-Roman VG, Mann DL, McNulty S, Semigran MJ, Lewis GD, de las Fuentes L, Joseph SM, Vader J, Hernandez AF, Redfield MM. Cardiovascular phenotype in HFpEF patients with or without diabetes: a RELAX trial ancillary study. J Am Coll Cardiol. 2014 Aug 12;64(6):541-9. doi: 10.1016/j.jacc.2014.05.030. PMID 25104521
- [Derived] Mohammed SF, Borlaug BA, McNulty S, Lewis GD, Lin G, Zakeri R, Semigran MJ, LeWinter M, Hernandez AF, Braunwald E, Redfield MM. Resting ventricular-vascular function and exercise capacity in heart failure with preserved ejection fraction: a RELAX trial ancillary study. Circ Heart Fail. 2014 Jul;7(4):580-9. doi: 10.1161/CIRCHEARTFAILURE.114.001192. Epub 2014 May 15. PMID 24833648
- [Derived] Zakeri R, Borlaug BA, McNulty SE, Mohammed SF, Lewis GD, Semigran MJ, Deswal A, LeWinter M, Hernandez AF, Braunwald E, Redfield MM. Impact of atrial fibrillation on exercise capacity in heart failure with preserved ejection fraction: a RELAX trial ancillary study. Circ Heart Fail. 2014 Jan;7(1):123-30. doi: 10.1161/CIRCHEARTFAILURE.113.000568. Epub 2013 Oct 25. PMID 24162898
- [Derived] Redfield MM, Borlaug BA, Lewis GD, Mohammed SF, Semigran MJ, Lewinter MM, Deswal A, Hernandez AF, Lee KL, Braunwald E; Heart Failure Clinical Research Network. PhosphdiesteRasE-5 Inhibition to Improve CLinical Status and EXercise Capacity in Diastolic Heart Failure (RELAX) trial: rationale and design. Circ Heart Fail. 2012 Sep 1;5(5):653-9. doi: 10.1161/CIRCHEARTFAILURE.112.969071. PMID 22991405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Sildenafil
Started | 103 | 113
Completed | 98 | 101
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Placebo; Sildenafil: 20 mg tid for 12 weeks followed by 60 mg tid for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Sildenafil | Total
Number analyzed (Participants) | 103 | 113 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 38 | 80
  >=65 years | 61 | 75 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (10.1) | 68.4 (10.5) | 68.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 48 | 64 | 112
Region of Enrollment [Number; unit: participants]
  United States | 93 | 101 | 194
  Canada | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Exercise Capacity, as Determined by Peak Oxygen Uptake
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 94 | 91
ml/min/kg | -0.07 (2.00) | -0.12 (2.29)

2. Secondary Outcome: Exercise Capacity, as Determined by Peak Oxygen Uptake
Time Frame: Change from Baseline to Week 12
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 96 | 97
ml/min/kg | 0.02 (1.70) | 0.03 (2.20)

3. Secondary Outcome: Exercise Capacity as Determined by Walk Distance
Description: 6 Minute Walk Distance
Time Frame: Change from Baseline to Week 12
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 96 | 99
meters | 26.2 (83.7) | 5.2 (69.1)

4. Secondary Outcome: Composite Score Reflective of Clinical Status
Description: Participants ranked sequentially with ranking stratified in one of three tiers based on:
  1. Death (lowest tier) The person with the shortest time from randomization to death is given the lowest rank within the tier.
  2. Hospitalizations due to cardiovascular or renal causes (middle tier) For patients alive, the ranking within this tier is based on time to hospitalization from randomization date. The person with the first cardiovascular or renal cause hospitalization will be given the lowest rank within the tier.
  3. Change in Minnesota Living with Heart Failure Questionnaire (MLWHFQ) from baseline (highest tier)
  The use of three tiers within the ranking reflects the greater adverse impact of death or cardiovascular hospitalization on clinical status without an arbitrary assignment as to the relative value of these events in relation to changes in quality of life. Rank order: 1-189 (higher values are better)
Time Frame: Measured at Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 94 | 95
units on a scale | 95.8 (55.0) | 94.2 (54.6)

5. Secondary Outcome: Exercise Capacity as Determined by Walk Distance
Description: 6 minute walk distance
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 90
meters | 17.5 (88.6) | 12.0 (94.2)

6. Secondary Outcome: Cardiopulmonary Exercise Test (CPET) Duration
Description: To interpret the CPET Exercise Duration change endpoints, an increase in exercise duration between Baseline and Week 12/Week 24 is considered to be an improvement
Time Frame: Change from Baseline to Week 12
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 91 | 88
minutes | 0.25 (1.61) | -0.15 (1.60)

7. Secondary Outcome: Cardiopulmonary Exercise Test (CPET) Duration
Description: as for outcome 6
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 89 | 86
minutes | 9.82 (2.63) | 9.77 (3.21)

8. Secondary Outcome: Ventilatory Anaerobic Threshold
Description: To interpret the Ventilatory Anaerobic Threshold (VAT) change endpoints, an increase in VAT between Baseline and Week 12/Week 24 is considered to be an improvement
Time Frame: Change from Baseline to Week 12
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 96 | 92
ml/min/kg | -0.01 (1.14) | 0.06 (1.24)

9. Secondary Outcome: Ventilatory Anaerobic Threshold
Description: as for outcome 8
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 94 | 88
ml/min/kg | -0.10 (1.26) | 0.17 (1.26)

10. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire (MLWHFQ)
Description: The MLWHFQ is a self-administered, disease-specific measure of health related quality of life (QOL) that assesses patients perceptions of the influence of heart failure on physical, socioeconomic and psychological aspects of life. Patients respond to 21 items using a six-point response scale (0-5). The total summary score can range from 0-105 with a lower score reflecting better heart failure related QOL. Two sub-scale scores reflect physical (8 items) and emotional (5 items) impairment.
  Total score: 0 - 105 Physical subscore: 0 - 40 Emotional subscore: 0 - 25
Time Frame: Change from Baseline to Week 12
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 97 | 95
units on a scale | -8.3 (22.0) | -6.2 (20.8)

11. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire
Description: The MLWHFQ is a self-administered, disease-specific measure of health related quality of life (QOL) that assesses patients perceptions of the influence of heart failure on physical, socioeconomic and psychological aspects of life. Patients respond to 21 items using a six-point response scale (0-5). The total summary score can range from 0-105 with a lower score reflecting better heart failure related QOL. Two sub-scale scores reflect physical (8 items) and emotional (5 items) impairment.
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 91 | 91
units on a scale | -9.2 (24.2) | -8.3 (19.7)

12. Other Pre Specified Outcome: MRI Left Ventricular Mass
Description: A decrease in LV Mass is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 47 | 49
gm | 0.29 (14.43) | -0.07 (14.93)

13. Other Pre Specified Outcome: MRI Left Ventricular Mass Index
Description: A decrease in Left Ventricular Mass Index is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: gm/m^2
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 47 | 49
gm/m^2 | 0.47 (6.54) | 0.61 (6.96)

14. Other Pre Specified Outcome: MRI Left Ventricular End Diastolic Volume
Description: An increase in Left Ventricular End Diastolic Volume is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 103 | 113
mL | -3.70 (21.03) | 3.61 (25.02)

15. Other Pre Specified Outcome: MRI Left Ventricular End Diastolic Volume Index
Description: An increase in Left Ventricular End Diastolic Volume Index is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 47 | 49
mL/m^2 | -1.73 (9.45) | 2.11 (11.21)

16. Other Pre Specified Outcome: MRI Left Ventricular End Systolic Volume Index
Description: An increase in Left Ventricular End Systolic Volume Index is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 47 | 49
mL/m^2 | -0.82 (4.09) | 0.25 (6.12)

17. Other Pre Specified Outcome: MRI Left Ventricular Ejection Fraction (LVEF)
Description: An increase in LVEF is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: percentage of volume
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 47 | 49
percentage of volume | 0.55 (4.28) | 0.62 (4.88)

18. Other Pre Specified Outcome: Echocardiogram Left Ventricular Mass
Description: A decrease in Left Ventricular Mass is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 56 | 58
gm | -1.93 (47.36) | -8.79 (35.60)

19. Other Pre Specified Outcome: Medial Diastolic Elastance
Description: A decrease in Medial Diastolic Elastance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: (m/sec)/cc
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 72 | 68
(m/sec)/cc | -0.03 (0.11) | -0.01 (0.10)

20. Other Pre Specified Outcome: Lateral Diastolic Elastance
Description: A decrease in Lateral Diastolic Elastance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: (m/sec)/cc
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 67 | 67
(m/sec)/cc | -0.00 (0.09) | -0.01 (0.08)

21. Other Pre Specified Outcome: Medial Left Ventricular Relaxation
Description: An increase in Left Ventricular relaxation is considered to be an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 83 | 77
m/sec | 0.00 (0.02) | -0.00 (0.02)

22. Other Pre Specified Outcome: Lateral Left Ventricular Relaxation
Description: An increase in Left Ventricular relaxation is considered to be an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 78 | 74
m/sec | -0.00 (0.02) | -0.00 (0.02)

23. Other Pre Specified Outcome: Medial Filling Pressure
Description: A decrease in medial filling pressure is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 80 | 75
m/sec | -1.64 (6.83) | 0.33 (6.04)

24. Other Pre Specified Outcome: Lateral Filling Pressure
Description: A decrease in lateral filling pressure is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 75 | 72
m/sec | -0.44 (5.17) | -0.04 (5.68)

25. Other Pre Specified Outcome: ECHO Effective Arterial Elastance
Description: A decrease in Effective Arterial Elastance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: Farads-1
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 76 | 68
Farads-1 | 0.03 (0.46) | -0.07 (0.36)

26. Other Pre Specified Outcome: ECHO Systemic Vascular Resistance
Description: A decrease in Systemic Vascular Resistance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: Woods units
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 74 | 66
Woods units | 0.01 (0.46) | -0.01 (0.35)

27. Other Pre Specified Outcome: MRI Effective Arterial Elastance
Description: A decrease in Effective Arterial Elastance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: Farads-1
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 45 | 47
Farads-1 | 0.04 (0.44) | -0.15 (0.38)

28. Other Pre Specified Outcome: MRI Systemic Vascular Resistance
Description: A decrease in Systemic Vascular Resistance is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: Woods units
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 45 | 47
Woods units | 0.06 (0.57) | -0.10 (0.39)

29. Other Pre Specified Outcome: MRI Aortic Thickness
Description: A decrease in Aortic Thickness is considered an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 33 | 31
mm | 0.01 (0.17) | -0.03 (0.18)

30. Other Pre Specified Outcome: MRI Aortic Distensibility
Description: An increase in Aortic Distensibility is considered to be an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: cm^2*dyne-1
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 31 | 29
cm^2*dyne-1 | 0.12 (0.66) | 0.29 (1.13)

31. Other Pre Specified Outcome: ECHO Pulmonary Artery Systolic Pressure
Description: A decrease in Pulmonary Artery Systolic Pressure is considered to be an improvement
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 58 | 45
mmHg | -0.15 (12.43) | 0.32 (10.09)

32. Other Pre Specified Outcome: Best Available Creatinine
Description: Best available=local lab results only when core lab results not available
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 98 | 100
mg/dL | 0.02 (0.23) | 0.09 (0.29)

33. Other Pre Specified Outcome: Best Available Glomerular Filtration Rate (GFR)
Description: Best available=local lab results when core lab results not available
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 98 | 100
mL/min/1.73m^2 | -0.91 (15.02) | -3.27 (12.16)

34. Other Pre Specified Outcome: Cystatin C
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
mg/L | -0.01 (0.27) | 0.10 (0.29)

35. Other Pre Specified Outcome: Uric Acid
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 94 | 94
mg/dL | -0.11 (1.79) | 0.51 (1.80)

36. Other Pre Specified Outcome: N-terminal Pro B-type Natriuretic Peptide (NT Pro-BNP)
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 94 | 95
pg/mL | -50.52 (799.87) | 158.25 (538.85)

37. Other Pre Specified Outcome: Aldosterone
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
pg/mL | 7.04 (220.06) | 1.22 (213.47)

38. Other Pre Specified Outcome: High Sensitivity Troponin I
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 93
pg/mL | 3.88 (29.71) | 11.11 (62.49)

39. Other Pre Specified Outcome: Procollagen III N-terminal Peptide
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 93 | 95
ug/L | 0.58 (5.22) | 0.41 (3.90)

40. Other Pre Specified Outcome: Endothelin-1
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
pg/mL | 0.04 (1.51) | 0.49 (1.29)

41. Other Pre Specified Outcome: High Sensitivity C-Reactive Protein
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
mg/L | 0.36 (7.20) | 0.32 (5.49)

42. Other Pre Specified Outcome: Collagen Type I (CITP)
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
ug/L | -0.17 (4.03) | 5.61 (48.96)

43. Other Pre Specified Outcome: Cyclic Guanosine Monophosphate (cGMP)
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 95 | 95
pmol/mL | 1.28 (37.05) | 8.72 (30.22)

44. Other Pre Specified Outcome: Galectin 3
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 93 | 92
ng/mL | 1.10 (9.63) | 1.26 (7.71)

45. Other Pre Specified Outcome: Furosemide-Equivalent Dose
Time Frame: Change from Baseline to Week 24
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Sildenafil
Number analyzed (Participants) | 98 | 100
mg | -0.23 (35.44) | 7.27 (59.53)

ADVERSE EVENTS:
Arm/Group | Placebo | Sildenafil
Serious Adverse Events (participants affected / at risk) | 16/103 | 25/113
Other Adverse Events (participants affected / at risk) | 72/103 | 83/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Sildenafil (N=113)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 7 | 9
Cardiac Failure Acute (Cardiac disorders) | 3 | 2
Palpitations (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypertensive Emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Implant Site Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4
Pyelonephritis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Sildenafil (N=113)
Angina Pectoris (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 0
Atrial Flutter (Cardiac disorders) | 1 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 5
Palpitations (Cardiac disorders) | 4 | 5
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 9
Hot Flush (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 8
Perhipheral Coldness (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 0 | 1
Varicose Vein (Vascular disorders) | 0 | 1
Balance Disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 11 | 9
Dizziness Postural (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 27
Memory Impairment (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 0 | 1
Diarhea (Gastrointestinal disorders) | 14 | 14
Tinnitis (Ear and labyrinth disorders) | 4 | 3
Visual Impairment (Eye disorders) | 5 | 7
Non-Cardiac Chest Pain (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No